CLINICAL TRIAL: NCT02050321
Title: A Phase II Study of Vemurafenib Combined With Acitretin in Patients With Advanced Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical company pulled support for the trial.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1312167559
Record Dates: First submitted 2014-01-24; First posted 2014-01-30 (Estimated); Results first posted 2017-04-19 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Acitretin; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acitretin and Vemurafenib (Experimental): Vemurafenib is self-administered at a dose of 960 mg (four 240 mg tablets) twice daily. The first dose should be taken in the morning and the second dose should be taken in the evening approximately 12 hours later. Each dose can be taken with or without a meal. Acitretin will initially be dosed at 25 mg orally per day with dosing altered every two weeks with a 50 mg dose.
  Interventions: Drug: Acitretin; Drug: Vemurafenib

INTERVENTIONS:
Drug: Acitretin — A combination of Acitretin and Vemurafenib will be administered to determine if it reduces the incidence of biopsy-confirmed cSCC at 6 months
  Other Names: Soriatane
Drug: Vemurafenib — A combination of Acitretin and Vemurafenib will be administered to determine if it reduces the incidence of biopsy-confirmed cSCC at 6 months
  Other Names: Zelboraf

SUMMARY:
We propose to conduct a phase 2 study to assess whether the addition of acitretin to vemurafenib therapy is able to decrease the rate of cutaneous squamous cell carcinoma (cSCC) development, a known side effect of vemurafenib therapy, in patients with advanced melanoma. Further, we seek a preliminary assessment as to whether the addition of acitretin to vemurafenib enhances the clinical efficacy of this anti-melanoma agent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced melanoma.
* BRAF mutation detected by DNA sequencing of exon 15.
* Age 18 or older.
* ECOG Performance Status 0-2.
* Appropriate tumor imaging studies (i.e. CT scan chest, abdomen and pelvis or PET/CT scan) performed within 28 days of study registration.
* Patients with melanoma measurable by RECIST 1.1 criteria will be monitored using this system for evidence of disease response/progression.
* Patients with a known history of brain metastases must have a diagnostic quality MRI of the brain or contrasted CT scan of the head performed within 28 days prior to registration.
* Female patients of child bearing capacity must have had 2 negative urine or serum pregnancy tests with a sensitivity of at least 25 mIU/mL before receiving the initial acitretin prescription. The first test (a screening test) is obtained by the prescriber when the decision is made to pursue acitretin therapy. The second pregnancy test (a confirmation test) should be done during the first 5 days of the menstrual period immediately preceding the beginning of acitretin therapy. The second test will be need to be repeated if not performed within 14 days prior to registration.
* Willingness to use at least two forms of contraception during sexual intercourse, including at least one form of barrier contraception, for at least 30 days prior to receiving the first dose of acitretin AND during the study period, AND up to 3 years after receiving the last dose of acitretin.
* Patients must agree not to consume alcoholic beverages while receiving acitretin and for 2 months after cessation of therapy.
* Electrocardiogram with QTc <450 ms at baseline.
* Patients must be evaluated for the following within 14 days prior to registration:

  * leukocytes >3,000/mcL
  * absolute neutrophil count >1,500/mcL
  * platelets >100,000/mcL
  * Hemoglobin >9.0 g/dL
  * AST(SGOT)/ALT(SGPT) <2.5 X institutional upper limit of normal
  * Alkaline phosphatase <2.5 X institutional upper limit of normal
  * Total bilirubin <1.5 X institutional upper limit of normal
  * Renal function serum creatinine <1.5 mg/dL OR 1.5 x institutional normal; alternatively, creatinine clearance as assessed by 24-hour urine collection ≥60 ml/min
  * Total cholesterol < 239 mg/dL or < 6.1 mmol/L
  * LDL < 159 mg/d or < 4.1mmol/L
  * HDL > 40 mg/dL or >1.0 mmol/L
  * Serum triglycerides < 199 mg/dL or < 2.2 mmol/L
  * Potassium 3.5-5.5 mMol/L
  * Magnesium 1.7-2.6mg/dL
  * Calcium 8.5-10.6 mg/dL

Exclusion Criteria:

* Known hypersensitivity to vemurafenib, acitretin, or vitamin A analogues.
* Uncontrolled hypertension.
* Serious and uncontrolled hypertriglyceridemia.
* Uncontrolled coronary artery disease or active anginal symptoms.
* Uncontrolled brain metastases.
* Concomitant malignancies or previous malignancies within the last 5 years, with the exception of adequately treated basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or low-grade prostate cancer.
* Myocardial Infarction, Transient Ischemic Attack (TIA), Cerebrovascular Accident (CVA) or symptomatic Congestive Heart Failure (CHF) within 6 months of study registration.
* Corrected QTc interval >450ms at baseline, history of congenital long QT syndrome, or known and uncorrectable electrolyte abnormalities.
* History of organ or hematologic transplant.
* Underlying defined genetic syndrome based on individual or family history predisposing to high risk of non-melanoma or melanoma skin cancer as assessed by the treating Oncologist.
* Concurrent use of St John's Wort.
* Concurrent (or within 60 days prior to acitretin dosing) use of methotrexate or other tetracyclines, phenytoin, vitamin A supplements, Tegison (etretinate) or progestin-only oral contraceptives.
* Pregnant or nursing.
* Receipt of any other investigational agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Cranmer, MD, PhD, Principal Investigator — University of Arizona
Locations (1):
- University of Arizona Cancer Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Acitretin and Vemurafenib
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acitretin and Vemurafenib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [52 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Development of cSCC at 6 Months (Biopsy Confirmed).
Time Frame: 6 months post treatment
Population: Per the PI: There is no measurable or interpretable data for this study. Only two patients were enrolled before the study closed to accrual due to recent FDA approvals of drugs for melanoma.Patients were removed from protocol prior to reaching data points or the completing the study.
Arm/Group | Acitretin and Vemurafenib
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Adverse Events
Description: The study period during which all AEs must be reported begins after informed consent is obtained and initiation of study treatment and ends 30 days following the last administration of study treatment or study discontinuation/termination, whichever is earlier. All adverse events will be classified using either the MedDRA term or NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Baseline through 30 Days post Treatment
Population: Per the PI: Although there is no measurable or interpretable data for this study. One patient had higher than normal liver lab results and was removed from study treatment due to grade and severity. Patient safety was evaluated.
Measure: Count of Participants; unit: Participants
Arm/Group | Acitretin and Vemurafenib
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: SAEs were collected on Day 1 and Day 15 of each of the 3 cycles. End of Treatment or Early Term SAEs were collected 30 days after the last dose of study drug.
Arm/Group | Acitretin and Vemurafenib
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acitretin and Vemurafenib (N=2)
Respiatory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Elevated Liver Values (Hepatobiliary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes